CLINICAL TRIAL: NCT01732341
Title: APPOSITION V: Stentys Coronary Stent System Clinical Trial in Patients With Acute Myocardial Infarction
Brief Title: Stentys Coronary Stent System Clinical Trial in Patients With Acute Myocardial Infarction
Acronym: APPOSITION V
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to discontinue patient follow-up at 2 years.
Sponsor: Stentys (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STENTYS
Record Dates: First submitted 2012-11-02; First posted 2012-11-22 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2015-11

CONDITIONS: Acute Myocardial Infarction
Keywords: STEMI; BMS; Self-expanding stent
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STENTYS self-apposing stent (Experimental): Intervention to treat STEMI with the STENTYS self-apposing stent
  Interventions: Device: STENTYS self-apposing stent
- VISION balloon-expandable stent (Active Comparator): STEMI treatment with a VISION balloon-expandable stent
  Interventions: Device: VISION balloon-expandable stent

INTERVENTIONS:
Device: STENTYS self-apposing stent — Intervention to treat STEMI with the STENTYS self-apposing stent
  Arms: STENTYS self-apposing stent
Device: VISION balloon-expandable stent — STEMI treatment with a VISION balloon-expandable stent
  --------------------------------------------------------------------------------
  Arms: VISION balloon-expandable stent

SUMMARY:
This study will test compare the Stentys Stent with the Multi-Link Vision™ stent system (Abbott Vascular Inc.)in patients with a heart attack. It is expected that the Stentys stent is not worse than the Vision stent.

DETAILED DESCRIPTION:
Coronary artery disease continues to be the most common cause of morbidity and mortality in the occidental world. Treatment of coronary atherosclerotic disease has been significantly advanced by interventional cardiology, and in particular the advent of coronary arterial stents. In comparison to angioplasty alone, stents have reduced the incidence of angiographic as well as clinical restenosis, the recurrence of angina, the need for coronary arterial bypass graft (CABG) surgery, the need for repeat revascularization and the occurrence of major adverse cardiac events (MACE).However,problems remain due to failure to achieve optimal stent apposition and normal myocardial reperfusion. Early stent malapposition may be due to incomplete expansion or undersizing of balloon-expandable stents. Several studies have emphasized the importance of early malapposition in the setting of ST elevation MI, in which substantial thrombotic burden and the presence of diffuse vasoconstriction may be contributory. The Stentys Coronary Stent System includes a self-expanding bare metal (nitinol) stent on a rapid exchange (RX) delivery system. In view of the theoretical implications of malapposition, the self-expanding property may offer a potential benefit.

This study is designed to evaluate the safety and effectiveness of the Stentys Coronary Stent System in the treatment of de novo stenotic lesions in coronary arteries in patients undergoing primary revascularization due to AMI as compared to the Multi-Link Vision™ coronary stent system (Abbott Vascular Inc. The study is powered for non-inferiority of the Stentys Coronary Stent System compared to the Vision Stent System.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Subject ≥ 18 years old.
2. Subject experiencing clinical symptoms consistent with AMI of >30 min. in duration.
3. ST elevation ≥1 mm in ≥2 contiguous leads or new left bundle branch block, or true posterior MI with ST depression of ≥1 mm in ≥2 contiguous anterior leads.
4. Symptom duration is <12 hours prior to signing informed consent.
5. Subject should be in catheterization laboratory and procedure started within 2 hours of consent.
6. Patient provides written informed consent.
7. Patient agrees to all required follow-up procedures and visits.

Angiographic Inclusion Criteria

1. Based on coronary anatomy, PCI is indicated for the culprit lesion with anticipated use of stenting.
2. The vessel diameter is either known or expected to be 2.5-4.0mm, without excessive tortuosity or diffuse distal disease.
3. Lesion length ≥12mm and ≤ 23mm

   -

Exclusion Criteria:

General Exclusion Criteria

1. Currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
2. A previous coronary interventional procedure of any kind within 30 days prior to the procedure.
3. Female patients of childbearing potential known to be pregnant.
4. Patients undergoing cardiopulmonary resuscitation.
5. Cardiogenic shock (SBP <80 mmHg for >30 minutes, or requiring IV pressors or emergency IABP for hypotension).
6. The subject requires multivessel PCI at time of index procedure or any staged procedure of the target vessel within 9 months or any non-target vessel within 30 days post-procedure.
7. The target lesion requires treatment with a device other than PTCA prior to stent placement (such as, but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.). Thrombus aspiration may be used per operator discretion.
8. Attempted thrombolysis.
9. Co-morbid condition(s) that could limit the subject's ability to participate in the trial or to comply with follow-up requirements, or impact the scientific integrity of the trial.
10. Concurrent medical condition with a life expectancy of less than 12 months.
11. Known left ventricular ejection fraction (LVEF) < 25% at the most recent evaluation (prior to the index hospitalization).
12. History of cerebrovascular accident or transient ischemic attack in the last 6 months.
13. Active peptic ulcer or active gastrointestinal (GI) bleeding.
14. History of bleeding diathesis or coagulopathy or inability to accept blood transfusions.
15. Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, cobalt, nickel, or sensitivity to contrast media, which cannot be adequately pre-medicated.
16. Known serum creatinine level > 2.5 mg/dl, eGFR <30, or hemodialysis dependent.

Angiographic Exclusion Criteria

1. Unprotected left main coronary artery disease (obstruction greater than 60% in the left main coronary artery that is not protected by at least one non-obstructed bypass graft to the left anterior descending (LAD) or left circumflex (LCX) artery or a branch thereof).
2. Multi-vessel intervention required during the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure | 12 months.
  From date of randomization until the date of first documented TVF, assessed up to 12 months.

SECONDARY OUTCOMES:
Acute Stent Malapposition | Immediately after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, MD, Principal Investigator — Mount Sinai Hospital, New York NY; Maurice Buchbinder, MD, Principal Investigator — Fouyndation Cardiovascular Research, La Jolla, CA
Locations (3):
- United States (2):
  - Foundation Cardiovascular medicine, La Jolla, California
  - Mount Sinai Hospital, New York, New York
- AMC, Amsterdam, Netherlands

REFERENCES:
- [Derived] Grundeken MJ, Lu H, Mehran R, Cutlip DE, Leon MB, Yeung A, Koch KT, Montalescot G, van Geuns RJ, Spaargaren R, Buchbinder M. APPOSITION V: STENTYS coronary stent system clinical trial in subjects with ST-segment elevation myocardial infarction--rationale and design. Am Heart J. 2014 Nov;168(5):652-60. doi: 10.1016/j.ahj.2014.07.011. Epub 2014 Jul 24. PMID 25440792